CLINICAL TRIAL: NCT03414424
Title: Non-invasive Cervical Electrical Stimulation for SCI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bronx VA Medical Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, Noam Y. Harel, Principal Investigator, Bronx VA Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: HAR-17-017
Record Dates: First submitted 2018-01-16; First posted 2018-01-30 (Actual); Results first posted 2023-11-29 (Actual); Last update posted 2023-11-29 (Actual); Status verified 2023-11

CONDITIONS: Spinal Cord Injuries
Keywords: transcutaneous electric nerve stimulation; transcranial magnetic stimulation
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- All subjects (Experimental): All subjects undergo same full protocol, including CES at rest and CES plus active hand or wrist movements.
  Interventions: Device: CES at rest; Device: CES plus active hand or wrist movements

INTERVENTIONS:
Device: CES at rest — CES will be delivered at rest at various intensities, in combination with either electrical stimulation over peripheral nerves or magnetic stimulation over the motor cortex.
  This is an experiment designed to measure CES interactions with other central and peripheral nerve circuits.
Device: CES plus active hand or wrist movements — CES will be delivered while the participant performs specific finger or wrist tasks at different degrees of effort.
  This is an experiment designed to detect momentary changes in muscle function.

SUMMARY:
Most spinal cord injuries (SCI) are anatomically incomplete - some nerve circuits remain intact, even if the individual cannot feel or control them. Activating spared nerve circuits may improve functional recovery.

With this goal, the Investigators have developed a form of electrical stimulation over the cervical spinal cord that can activate muscles in both hands simultaneously and comfortably. This technique, called cervical electrical stimulation (CES), works at the skin surface - no surgery or other invasive procedures are required.

The long-term goal is to use CES to strengthen residual circuits to hand muscles after SCI. Regaining control over hand function represents the top priority for individuals with cervical SCI.

In the current study, the Investigators first need to better understand how CES works. In the first half of this study, the Investigators will take a systematic approach to determining how CES interacts with other circuits in the spinal cord and the brain. In the second half of the study, the Investigators will test combinations of CES with active hand and wrist movements to find ways to enhance physical movement with CES.

These experiments will improve understanding of electrical stimulation in SCI, and may set the table for future treatments to prolong any short-term benefits observed in this study.

DETAILED DESCRIPTION:
Roughly 60% of spinal cord injuries occur at the cervical level. Most injuries are anatomically incomplete. Activating spared nerve circuits augments functional recovery of the damaged nervous system. With this goal, the Investigators have developed a novel method of non-invasive cervical electrical stimulation (CES). Preliminary data show that CES triggers afferent sensory or efferent motor nerve roots depending on stimulus intensity, resulting in concurrent activation of multiple muscles on both upper limbs. the Investigators aim to use CES to strengthen residual circuits to hand muscles after SCI. Regaining control over hand function represents the top priority for individuals with cervical SCI.

However, much more work needs to be done to better understand underlying CES mechanisms, its interactions with segmental and supraspinal circuits, and its optimal stimulation parameters for improving neural transmission to the hands. This proposal will address these issues.

Mechanistic experiments: 15 able-bodied volunteers and 15 subjects with motor-incomplete cervical spinal cord injury will undergo systematic combinations of CES with transcranial magnetic stimulation (TMS) or peripheral nerve stimuli at varying intensities, sites, and interstimulus intervals.

Mechanistic hypotheses: Conditioning subthreshold CES pulses will potentiate responses to test pulses of TMS and peripheral nerve F-wave stimulation, will reduce responses to test pulses of peripheral nerve H-reflex stimulation, and will modulate response to test suprathreshold CES pulses in either direction depending on conditioning stimulus interval and intensity. These experiments will elucidate CES circuit interactions at both the segmental and supraspinal levels.

Combined CES-volitional movement experiments: 15 able-bodied volunteers and 15 subjects with motor-incomplete cervical spinal cord injury will undergo systematic combinations of CES with volitional wrist and hand movements at varying intensity and effort level.

Combined CES-volitional movement hypotheses: Conditioning subthreshold CES pulses will facilitate concurrent volitional wrist and hand muscle activation. Suprathreshold CES will transiently inhibit concurrent volitional wrist and hand muscle activation. These experiments will shed light on the clinically relevant possibility of using CES to enhance response to physical exercise therapy.

Completion of the proposed studies will characterize CES circuit timing and distribution, and will demonstrate in principle the potential for CES to enhance physical therapy for wrist and hand muscles. Furthermore, this approach is compatible with other interventions, including drug and cell-based treatments.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 75 years;
* Chronic (more than 12 months since injury) incomplete SCI between levels C2-C8.
* Incomplete weakness of left or right hand muscles: score of 2, 3, or 4 (out of 5) on manual muscle testing of finger extension, finger flexion, or finger abduction;
* Detectable F-wave responses of the left or right abductor pollicis brevis muscle to median nerve stimulation.
* US Veteran or non-Veteran

Exclusion Criteria:

* History of other serious injury or disease of central or peripheral nervous system
* History of seizures
* Ventilator dependence or patent tracheostomy site
* Use of medications that significantly lower seizure threshold
* History of head trauma with evidence of brain contusion or hemorrhage or depressed skull fracture on prior imaging
* History of implanted:

  * brain/spine/nerve stimulators
  * aneurysm clips
  * ferromagnetic metallic implants
  * or cardiac pacemaker/defibrillator
* Significant coronary artery or cardiac conduction disease
* Recent history (within past 6 months) of recurrent autonomic dysreflexia, defined as a syndrome of sudden rise in systolic pressure greater than 20 mm Hg (millimeters of mercury) or diastolic pressure greater than 10 mm Hg, without rise in heart rate, accompanied by symptoms such as headache, facial flushing, sweating, nasal congestion, and blurry vision (this will be closely monitored during all screening and testing procedures);
* History of bipolar disorder or suicide attempt or active psychosis
* Heavy alcohol consumption (> equivalent of 5 ounces of liquor) within previous 48 hours
* Open skin lesions over the face, neck, shoulders, or arms
* Pregnancy
* Unsuitable for study participation as determined by study physician

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2017-08-22 (Actual); Primary Completion 2021-04-30 (Actual); Study Completion 2021-04-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Noam Y. Harel, MD, PhD, Principal Investigator — Bronx VA Medical Center
Locations (1):
- James J. Peters VA Medical Center, Bronx, NY, The Bronx, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
A Limited Dataset (LDS), with individual electrophysiological and physiological outcome measures, will be shared in electronic format pursuant to a VA-approved Data Use Agreement. Individually Identifiable Data will be shared pursuant to valid HIPAA Authorization, Informed Consent, and an appropriate written agreement limiting use of the data to the conditions as described in the authorization and consent, and a written assurance from the recipient that the information will be maintained in accordance with the security requirements of 38 CFR Part 1.466.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: At time of publication
Access Criteria: A Limited Dataset (LDS) will be shared in electronic format pursuant to a VA-approved Data Use Agreement. Individually Identifiable Data will be shared pursuant to valid HIPAA Authorization, Informed Consent, and an appropriate written agreement limiting use of the data to the conditions as described in the authorization and consent, and a written assurance from the recipient that the information will be maintained in accordance with the security requirements of 38 CFR Part 1.466.

REFERENCES:
- [Background] Wu YK, Levine JM, Wecht JR, Maher MT, LiMonta JM, Saeed S, Santiago TM, Bailey E, Kastuar S, Guber KS, Yung L, Weir JP, Carmel JB, Harel NY. Posteroanterior cervical transcutaneous spinal stimulation targets ventral and dorsal nerve roots. Clin Neurophysiol. 2020 Feb;131(2):451-460. doi: 10.1016/j.clinph.2019.11.056. Epub 2019 Dec 13. PMID 31887616
- [Result] Wecht JR, Savage WM, Famodimu GO, Mendez GA, Levine JM, Maher MT, Weir JP, Wecht JM, Carmel JB, Wu YK, Harel NY. Posteroanterior Cervical Transcutaneous Spinal Cord Stimulation: Interactions with Cortical and Peripheral Nerve Stimulation. J Clin Med. 2021 Nov 15;10(22):5304. doi: 10.3390/jcm10225304. PMID 34830584

RESULTS

PARTICIPANT FLOW:
Groups:
- Able Bodied; Spinal Cord Injured: All subjects undergo same full protocol, including CES at rest and CES plus active hand or wrist movements.
  CES at rest: CES will be delivered at rest at various intensities, in combination with either electrical stimulation over peripheral nerves or magnetic stimulation over the motor cortex.
  This is an experiment designed to measure CES interactions with other central and peripheral nerve circuits.
  CES plus active hand or wrist movements: CES will be delivered while the participant performs specific finger or wrist tasks at different degrees of effort.
  This is an experiment designed to detect momentary changes in muscle function.
Period: Overall Study
Arm/Group | Able Bodied | Spinal Cord Injured
Started | 15 | 15
Completed | 15 | 12
Not Completed | 0 | 3
Not completed — Screened out after consent | 0 | 2
Not completed — Lost to Follow-up | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Able Bodied | Spinal Cord Injured | Total
Number analyzed (Participants) | 15 | 15 | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.7 (15.0) | 47.5 (15.4) | 43.1 (15.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 4 | 7
  Male | 12 | 11 | 23
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 2 | 4
  Not Hispanic or Latino | 11 | 12 | 23
  Unknown or Not Reported | 2 | 1 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 2 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 7 | 2 | 9
  White | 6 | 10 | 16
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 1 | 3
Region of Enrollment [Number; unit: participants]
  United States | 15 | 15 | 30

OUTCOME MEASURES:

1. Primary Outcome: Electromyographic Responses (Active)
Description: Effect of cervical electrical stimulation (CES) on concurrent finger or wrist active movements will be measured via root-mean-square of ongoing muscle activity in various hand and forearm muscles.
Time Frame: up to one day
Population: Data collection for this outcome was plagued with technical problems. The relative timing of cervical stimulation relative to active effort was irregularly applied. Grant funding expired.
  It is not possible to analyze the data collected for this aim.
Groups:
- Able-bodied: Volunteers without spinal cord injury.
- Spinal Cord Injury: Participants with chronic SCI between levels C2-C8
Arm/Group | Able-bodied | Spinal Cord Injury
Number analyzed (Participants) | 0 | 0

2. Primary Outcome: Electromyographic Responses to Transcranial Magnetic and Cervical Electrical Stimulation at Rest
Description: Response of the target hand muscle to transcranial magnetic stimulation (delivered at 120% of resting motor threshold) with or without a conditioning cervical electrical stimulator pulse (delivered at 90% of resting motor threshold) timed to arrive at cervical synapses 2 milliseconds after transcranial pulse arrival. Response is expressed as percentage change relative to the response to unconditioned transcranial magnetic stimulation.
Time Frame: up to one day
Population: Two enrolled spinal cord injury (SCI) participants failed screening. Data for transcranial magnetic stimulation (TMS) were excluded from two more SCI participants who were found after screening to either have unacceptable electrical background electromyographic activity or unreliable responses in resting muscle during TMS.
Measure: Mean (Standard Error); unit: % change from unconditioned TMS.
Arm/Group | Able-bodied | Spinal Cord Injury
Number analyzed (Participants) | 15 | 11
% change from unconditioned TMS. | 6.1 (8.9) | 32.0 (27.8)

ADVERSE EVENTS:
Time Frame: 1 week
Arm/Group | Able-bodied | Spinal Cord Injury
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/15
Other Adverse Events (participants affected / at risk) | 7/15 | 7/15
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Able-bodied (N=15) | Spinal Cord Injury (N=15)
Scalp pain/Headache (Nervous system disorders) | 3 | 3
Neck pain (Musculoskeletal and connective tissue disorders) | 2 | 3
Sleepy (General disorders) | 0 | 1
Depressed mood (Psychiatric disorders) | 1 | 0 — Temporary
Paresthesias (Nervous system disorders) | 1 | 0
Light-headed (General disorders) | 0 | 1
Metallic taste (Nervous system disorders) | 2 | 0
Trouble concentrating (Psychiatric disorders) | 2 | 0 — Transient

LIMITATIONS AND CAVEATS:
Data collection for the active condition (cervical electrical stimulation during active muscle contraction) was plagued with technical problems, not possible to quantitatively analyze.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-12-09): https://cdn.clinicaltrials.gov/large-docs/24/NCT03414424/Prot_SAP_001.pdf